CLINICAL TRIAL: NCT00026429
Title: A Multicenter Phase II Evaluation Of ONTAK (DENILEUKINDIFTITOX) In Patients With Low Or Intermediate Grade-B-Cell Non-Hodgkin's Lymphoma Who Have Been Treated Previously With A Monoclonal Antibody Or Who Are Not Candidates For Monoclonal Antibody Therapy
Brief Title: Denileukin Diftitox in Treating Patients With Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pharmatech Oncology (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069029; PHARMATECH-LP-ONT-BL; LIGAND-PHARMATECH-LP-ONT-BL; PHARMATECH-20002024
Record Dates: First submitted 2001-11-09; First posted 2004-02-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2002-02

CONDITIONS: Leukemia; Lymphoma
Keywords: stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — denileukin diftitox

INTERVENTIONS:
Biological: denileukin diftitox

SUMMARY:
RATIONALE: Biological therapies such as denileukin diftitox may be able to deliver cancer-killing substances directly to non-Hodgkin's lymphoma cells.

PURPOSE: Phase II trial to study the effectiveness of denileukin diftitox in treating patients who have non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of denileukin diftitox in patients with stages I-IV low- or intermediate-grade B-cell non-Hodgkin's lymphoma. II. Determine the safety of this drug in these patients.

OUTLINE: This is a multicenter study. Patients receive denileukin diftitox IV over 30-60 minutes on days 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients may receive up to 2 additional courses after achieving complete response. Patients are followed every 3 months until they have progressed or for 2 years from date of termination.

PROJECTED ACCRUAL: A total of 58 patients (29 with low-grade non-Hodgkin's lymphoma (NHL) and 29 with intermediate-grade NHL) will be accrued for this study within 12 months. The study may be stopped after accrual of 20 patients (10 with low-grade NHL and 10 with intermediate-grade NHL) if observed response rate is less than 1 in 10 for each stratum.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed low-grade B-cell non-Hodgkin's lymphoma (NHL) Working Formulation classification: Small lymphocytic lymphoma Follicular lymphoma (small cleaved or mixed small and large cell) REAL classification: B-cell chronic lymphocytic leukemia/small lymphocytic Lymphoplasmacytoid Marginal zone/MALT Follicular small or mixed small and large cell OR Histologically confirmed intermediate-grade B-cell NHL Working Formulation classification: Follicular large cell Diffuse small cleaved cell Diffuse mixed small and large cell Diffuse large cell REAL classification: Mantle cell Diffuse small cell Marginal zone/MALT Large B-cell Lymphoplasmacytoid Stage I, II, III, or IV disease No cutaneous T-cell lymphoma or other T-cell NHL Bidimensionally measurable disease Unidimensionally measurable disease allowed for mediastinal lymphoma only if outside previously irradiated field or there is evidence of progression Received prior monoclonal antibody therapy OR ineligible for monoclonal antibody therapy A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,000/mm3 Platelet count at least 50,000/mm3 Hemoglobin at least 8 g/dL Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) AST and ALT no greater than 1.5 times ULN Albumin at least 3.0 g/dL No chronic hepatitis Renal: Creatinine less than 1.8 mg/dL Cardiovascular: No New York Heart Association class III or IV heart disease No poorly controlled hypertension Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception HIV negative No serious concurrent illness or active infection requiring parenteral antibiotics that would preclude study No known hypersensitivity to study drug or its components, including diphtheria toxin, interleukin-2, or excipients No other malignancy within the past 5 years except resected basal or squamous cell skin cancer or carcinoma in situ of the cervix (prostate cancer in situ or breast cancer in situ within the past 5 years is allowed if patients are in complete remission with no active disease, have stable tumor markers for at least 3 months, and have a life expectancy of at least 2 years)

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Prior bone marrow transplantation allowed No prior denileukin diftitox or DAB486 IL-2 No concurrent immunotherapy Chemotherapy: No concurrent chemotherapy Endocrine therapy: No concurrent hormonal anticancer therapy Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy No prior radiotherapy to sole site of disease unless evidence of progression No concurrent radiotherapy Surgery: Not specified Other: At least 1 month since prior investigational agent No other concurrent experimental medications, including approved drugs tested in an investigational setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-01

CONTACTS AND LOCATIONS:
Overall Officials: Debby Henkens, Study Chair — Pharmatech Oncology
Locations (6):
- United States (6):
  - ION/Pharmatech Network, Pomona, California
  - Cancer and Blood Institute of the Desert, Rancho Mirage, California
  - Missouri Cancer Care, P.C., Saint Charles, Missouri
  - Nassau Hematology/Oncology PC, Lake Success, New York
  - Coastal Cancer Center, Myrtle Beach, South Carolina
  - Boston Baskin Cancer Group, University Tennessee Oncology/Hematology Group, Memphis, Tennessee